CLINICAL TRIAL: NCT00267410
Title: Adopting and Demonstrating the Adaptation of Prevention Techniques (ADAPT), Harlem United Community AIDS Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-CGH-4869; CA 2 U65/CCU223844-0101
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Sexually Transmitted Diseases; HIV Infections
Keywords: HIV; Adaptation; Behavioral interventions; Seropositive; MSM; HIV Seronegativity
MeSH Terms: conditions — Sexually Transmitted Diseases; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Healthy Relationships — "Healthy Relationships," grounded in the social cognitive theory, is a five-session, group-level intervention originally designed for HIV-positive heterosexual individuals seeking skills-building and support around risk reduction, as well as disclosure of status and sexual preference. Through clip media and active role-plays, the intervention promotes the development of decision-making and problem-solving tools, empowering participants to make voluntary and informed decisions around disclosure and safer sex practices. This model was formally disseminated to AIDS Service Organizations as part of CDC's strategic plan - Advancing HIV Prevention, New Strategies for a Changing Epidemic - which focused on innovative strategies to recruit individuals into HIV testing, as well as a movement towards secondary prevention efforts.

SUMMARY:
This project will pilot test a step-by-step guide for community-based organizations to engage in evidence-based adaptation of interventions previously shown to be effective in research settings for use in real world applications. The main purpose of this program is to improve understanding of the processes needed for adapting evidence-based behavioral interventions to fit new conditions or populations and to pilot CDC-developed draft guidance for adaptation. The second purpose of the program is to increase the number of effective behavioral HIV prevention interventions for 18-24 year old sero-positive men of color who have sex with other men (MSM of color).

DETAILED DESCRIPTION:
The Adopting and Demonstrating the Adaptation of Prevention Techniques project (referred to as ADAPTATION throughout this protocol) responds to concerns from the field that existing interventions do not address the HIV prevention needs of diverse and often unstudied populations. This project will pilot test a step-by-step guide for community-based organizations to engage in evidence-based adaptation of interventions previously shown to be effective in research settings for use in real world applications. The main purpose of this program is to improve understanding of the processes needed for adapting evidence-based behavioral interventions to fit new conditions or populations and to pilot CDC-developed draft guidance for adaptation. The second purpose of the program is to increase the number of effective behavioral HIV prevention interventions for 18-24 year old sero-positive men of color who have sex with other men (MSM of color).

Harlem United Community AIDS Center is one of five sites originally funded through Program Announcement 04064 and selected to receive a supplement to conduct adaptation activities. Under Program Announcement 04064, Harlem United, a community-based organization with over 16 years of experience providing quality HIV services to the Harlem and South Bronx communities, was funded to implement a multi-faceted, HIV prevention program. The program combines rapid testing, access to care, and an evidenced-based, group-level behavioral intervention (i.e., Healthy Relationships) for sero-positive, heterosexual men and women of color. Healthy Relationships is a five-session, small group-level intervention for persons living with HIV/AIDS that promotes the development of decision-making and problem-solving skills that enable participants to make informed and safe decisions about disclosure and behaviors. Preliminary evaluation efforts suggest that this service model is effective in reducing risk behaviors among the general population, but its appropriateness and effectiveness for specific sub-populations has yet to be fully demonstrated. The original research for Healthy Relationships was conducted in Atlanta, Georgia. Approximately half of the participants identified as gay and the study population had a mean age of 40 years. Harlem United will adapt the Healthy Relationships intervention for young sero-positive MSM of color between the ages of 18-24 who reside in Harlem, New York. Further adaptation also may include adding decision-making for disclosure with needle sharing partners.

The goal of Harlem United's ADAPTATION project is to evaluate efforts to adapt and implement the Healthy Relationships intervention for young sero-positive MSM of color by: 1) documenting the resources and activities required to adapt and implement the Healthy Relationships intervention model for young sero-positive MSM of color; 2) optimizing service delivery; 3) measuring the effectiveness of the newly-adapted intervention; and 4) assessing CDC's guidance for adapting effective behavioral interventions for new populations.

ELIGIBILITY:
Inclusion Criteria:

* MSM, at least 18 years old;
* HIV-positive; and
* Self-identified African Americans, English speaking African-born individuals and Latinos.

Exclusion Criteria:

* Non-English speaking;
* Under 18 years of age;
* Serious mental illness which makes them unsuitable for interviewing (accommodation will be made for HIV-related cognitive deficits & related illnesses);
* Inebriated;
* Has been interviewed before; and
* Anyone who does not meet the inclusion criteria.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2005-11; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Document the resources and activities required to adapt and implement the Healthy Relationships intervention model for young sero-positive MSM of color | 11/2005-9/2007
Measure the effectiveness of the newly-adapted intervention | 11/2005-9/2009
Assess CDC's guidance for adapting effective behavioral interventions for new populations. | 11/2005-11/2007

SECONDARY OUTCOMES:
Optimize service delivery | 11/2005-12/2009

CONTACTS AND LOCATIONS:
Overall Officials: Soraya Elcock, Principal Investigator — Harlem United Community AIDS Center
Locations (1):
- Harlem United Community AIDS Center, New York, New York, United States